CLINICAL TRIAL: NCT06185738
Title: WeCanManage: An mHealth Self-management Tool to Empower Survivors With Disabilities Due to Long-term Effects of Cancer and Its Treatment
Brief Title: WeCanManage. An mHealth Self-management Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Northwestern University (Other); Northeastern Illinois University (Other)
Responsible Party: Principal Investigator, Susan Magasi, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-1067
Record Dates: First submitted 2023-12-15; First posted 2023-12-29 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Head and Neck Cancer; Sarcoma
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Sarcoma

STUDY DESIGN:
Intervention Model Description: All participants will have a data collection session by phone lasting about 60 minutes, and to complete a demographic and health questionnaire, that includes questions such as sex, age, race, ethnicity, marital status, cancer type, time since diagnosis, date of diagnosis, stage of illness, type of primary treatment, type of disability, current activity level, health conditions, annual income, educational history.
  WeCanManage (WCM) app orientation by Zoom lasting about 60 minutes. Participants will complete WCM app program, about 10 minutes per day for 30 days and up to 45 days. Data collection by phone lasting about 60 minutes after completion of WCM app program and 4 weeks after completion of WCM app program All participants will have an intervention of 4 modules (WeCanRelate, WeCanAdapt, WeCanBe, and WeCanSpeakUp) that are presented as series of micro-learning sessions
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WCM app (Other): WCM app evaluation at baseline, upon completion of WCM program and 4 weeks after completion of WCM program, by completing PROMIS and Self Efficacy for managing disease scale questionnaires
  Interventions: Other: WCM app

INTERVENTIONS:
Other: WCM app — WCM app evaluation at baseline, at completion of WCM program and 4 weeks after completion of WCM program, by completing PROMIS and Self Efficacy for managing disease scale questionnaires

SUMMARY:
Examine the Feasibility, Acceptability, User Satisfaction, and Response Patterns and Preliminary Efficacy on Targeted Patient Reported Outcomes. Using a pre-post, single arm feasibility design with cancer survivors with disabilities

DETAILED DESCRIPTION:
Examine the Feasibility, Acceptability, User Satisfaction, and Response Patterns and Preliminary Efficacy on Targeted Patient Reported Outcomes. Using a pre-post, single arm feasibility design with cancer survivors with disabilities, we will collect data on the WeCanManage app delivered self-management intervention's feasibility, acceptability, user satisfaction as well as response patterns and preliminary efficacy on targeted patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

Usability Testing of the WeCanManage High Fidelity Prototype

* Age 18 or older
* Diagnosis of breast cancer, head and neck cancer or sarcoma
* Completion of active treatment
* Self-identify as a person with a disability according to the Americans with Disabilities .Act and the American Community Survey 6-disability questions
* Able to understand and communicate in English
* Medically stable enough to participate in two data collection sessions totaling 2 hours

Evaluation of the WeCanManage App

* Age 18 or older
* Diagnosis of breast cancer, head and neck cancer or sarcoma
* Completion of primary (i.e. surgery, chemotherapy, and/or radiation); may still be under-going endocrine or hormone therapies
* Self-identify as experiencing disabling after-effects of cancer and its treatment according to the Americans with Disabilities Act and the American Community Survey 6-disability questions
* Able to read, understand and communicate in English
* Ownership of a smartphone, tablet, or personal computer.
* Internet access

Exclusion Criteria:

Usability Testing of the WeCanManage High Fidelity Prototype

* No diagnosis of breast cancer, head and neck cancer or sarcoma
* In active treatment
* Does not self-identify as a person with a disability according to the Americans with Disabilities Act and the American Community Survey 6-disability questions
* Not able to understand and communicate in English
* Not medically stable enough to participate in two data collection sessions totaling 2 hours

Evaluation of the WeCanManage App

* Age 17 or younger
* No diagnosis of breast cancer, head and neck cancer or sarcoma
* In active treatment
* Does not self-identify as experiencing long-term effects of cancer and its treatment according to the Americans with Disabilities Act and the American Community Survey 6-disability questions
* Not able to read, understand, and communicate in English
* Does not have access to internet enabled smartphone, tablet, or personal computer
* Does not have access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of WCM app | 1 year
  Evaluate recruitment capability by assessing response rate
Feasibility of WCM app | 1 year
  Number of participants that started the intervention from consent
Acceptability of WCM app | 1 year
  Number of participants that adhered to the intervention
Acceptability of WCM app | 1 year
  Number of participants that were engaged in the intervention
Acceptability of WCM app | 1 year
  Number of participants that were satisfied with the intervention
Acceptability of WCM app | 1 year
  Number of participants that found the intervention helpful
Acceptability of WCM app | 1 year
  Number of participants that wished to continue using the intervention l
Feasibility with WCM app | Baseline
  Measurement of PROMIS questionnaire, low score health good, high score health not good
Feasibility with WCM app | 4 Weeks
  Measurement of PROMIS questionnaire, low score health good, high score health not good
Feasibility with WCM app | 8 Weeks
  Measurement of PROMIS questionnaire, low score health good, high score health not good
Feasibility with WCM app | Baseline
  Measurement of Self Efficacy for managing disease scale questionnaire, low score not confident, high score very confident
Feasibility with WCM app | 4 weeks
  Measurement of Self Efficacy for managing disease scale questionnaire, low score not confident, high score very confident
Feasibility with WCM app | 8 weeks
  Measurement of Self Efficacy for managing disease scale questionnaire, low score not confident, high score very confident

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois, Chicago, Illinois, United States